CLINICAL TRIAL: NCT06387459
Title: Safety and Feasibility of Knee Extensor Muscle-mimicking, Fabric-type Orthosis on Gait in Geriatric Patients: Pilot Clinical Trial
Brief Title: Feasibility of Fabric Orthosis for Knee Support in Elderly Gait Improvement
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Ministry of Science and ICT, Republic of Korea (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2022M3C1A3090827
Record Dates: First submitted 2024-04-22; First posted 2024-04-29 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2024-07

CONDITIONS: Gait; Fall; Orthotic Devices
Keywords: Geriatric patient

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Knee Extensor Muscle-Mimicking Orthosis (Experimental): This arm involves participants wearing a novel, lightweight fabric-type orthosis designed to mimic the function of knee extensor muscles through embedded shape-memory alloys. This intervention aims to support the knee joint during gait, enhancing stability and mobility for elderly individuals with compromised muscle function.
  Interventions: Device: Fabric-Type Knee Extensor Muscle-Mimicking Orthosis

INTERVENTIONS:
Device: Fabric-Type Knee Extensor Muscle-Mimicking Orthosis — The intervention device is a fabric-based orthosis incorporating shape-memory alloy springs designed to mimic the action of knee extensor muscles. The primary function of this orthosis is to provide supplementary support to the knee joint during walking, aiming to stabilize the gait of elderly individuals affected by muscle weakness or degenerative joint conditions. Material: The orthosis is made from a lightweight, flexible fabric that allows for breathability and comfort during extended wear. Mechanism: Embedded within the fabric are shape- memory alloy springs that function similarly to biological muscles.

SUMMARY:
This pilot clinical trial assesses the safety and feasibility of a novel fabric-type orthosis designed to mimic the knee extensor muscles and improve gait in elderly patients with mobility impairments due to conditions like sarcopenia, diabetes, or knee osteoarthritis. The study aims to test this orthosis in a real- world setting to see if it can enhance mobility and stability for elderly individuals, potentially reducing falls and improving quality of life. A total of 30 participants aged 65 and older will be recruited to use this orthosis across multiple sessions, where their gait will be analyzed under various conditions to measure the device's impact on walking speed, stability, and muscle activation.

DETAILED DESCRIPTION:
Objectives:

* Primary Objective: To evaluate the safety and feasibility of the fabric-type knee extensor muscle-mimicking orthosis in improving gait among elderly patients.
* Secondary Objectives: To measure changes in walking speed, endurance, and muscle activity to infer potential benefits in daily mobility.

Study Design:

* Study Population: 30 elderly patients suffering from conditions affecting mobility (sarcopenia, diabetes, knee osteoarthritis).
* Intervention: Use of a fabric-type orthosis mimicking knee extensor function, equipped with shape-memory alloy for dynamic movement support.
* Methodology:

  1. Training and Adaptation: Participants will undergo an initial training session to get accustomed to the orthosis, including donning and doffing, adjustment, and use in various environments (flat surfaces, inclines).
  2. Assessment Protocol:
* Before wearing the orthosis-after wearing the orthosis (power off)-after wearing the orthosis (power on)
* Walking environment will include EMG (Electromyography) measurements, 6-minute walk test, 10-meter walk test, and comprehensive gait analysis using platforms like the GAITRite system.
* Seating environment will include EMG (Electromyography) measurements and TUG test. 3. Safety Monitoring: Continuous monitoring of physiological responses (blood pressure, heart rate), musculoskeletal assessments, and skin integrity checks to monitor for adverse reactions or discomfort

ELIGIBILITY:
Inclusion Criteria:

Eligibility for participation in the study requires that all the following criteria are met:

1. Age: Participants must be 65 years of age or older.
2. Comprehension and Compliance: Able to fully understand and comply with the instructions and study procedures.
3. Mobility-Impacting Conditions: Must have at least one of the following conditions affecting mobility: (1)Sarcopenia:

   * Muscle Strength: Handgrip strength of <28 kg for men and <18 kg for women.
   * Muscle Function: Short Physical Performance Battery (SPPB) score of 8 or less.
   * Muscle Mass: Bioelectrical impedance analysis (BIA) showing muscle mass <7.0 kg/m² for men and <5.7 kg/m² for women. (2)Diabetes:
   * Diagnosed distal symmetric polyneuropathy.
   * Sensory impairments in toes or feet. (3)Knee Osteoarthritis:
   * Kellgren-Lawrence grade ≥2.
   * Persistent pain (≥3 months) with a severity of at least 3 on the Numerical Rating Scale (NRS).

Exclusion Criteria:

Individuals meeting any of the following criteria will be excluded from study participation:

1. Inability to Consent: Unable to provide informed consent or not willing to participate in the study procedures.
2. Severe Sensory or Motion Limitations: Including severe visual or vestibular impairments that could increase the risk of falling.
3. Communication Barriers: Significant hearing, speech, or language problems that would hinder communication with study personnel.
4. Independent Walking Inability: Cannot walk independently without the aid of a walking device.
5. Other Significant Diseases or Conditions:

   * Neurological disorders that affect walking ability (e.g., stroke, Parkinson's disease).
   * Orthopedic or musculoskeletal conditions severely affecting lower limb function.
   * Severe cardiovascular conditions including uncontrolled hypertension or heart failure.
   * Respiratory diseases requiring regular oxygen therapy.
   * Active cancer treatment or cancer treatment within the past 3 years (except basal cell carcinoma or localized prostate cancer).
   * Severe psychiatric disorders like schizophrenia or bipolar disorder.
6. Other Exclusionary Factors:

   * Past severe orthopedic surgeries on lower limbs which might affect gait and mobility.
   * Severe back pain or any other condition affecting mobility not already listed.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-07-31 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2026-05-14 (Estimated)

PRIMARY OUTCOMES:
Completion Rate | 1.Baseline (before brace application) 2.Immediately post-brace application (power off), 3.Immediately post-brace activation (power on)
  The proportion of participants who complete the study as per the protocol, which indicates the orthosis's acceptability and the study's overall manageability.

SECONDARY OUTCOMES:
Dropout Rate | 1.Baseline (before brace application) 2.Immediately post-brace application (power off), 3.Immediately post-brace activation (power on)
  Measures participant retention throughout the study, providing insights into the orthosis's usability and participant satisfaction.
User Feedback | 1.Baseline (before brace application) 2.Immediately post-brace application (power off), 3.Immediately post-brace activation (power on)
  Collected using the Quebec User Evaluation of Satisfaction with assistive Technology 2.0 (QUEST 2.0), which will cover aspects such as the orthosis's comfort, ease of use, safety, and effectiveness. This feedback is vital for understanding user satisfaction and for guiding future improvements.
6-Minute Walk Test | 1.Baseline (before brace application) 2.Immediately post-brace application (power off), 3.Immediately post-brace activation (power on)
  To measure the distance covered in six minutes as a test of aerobic capacity and endurance, which may improve with the use of the orthosis.
10-Meter Walk Test | 1.Baseline (before brace application) 2.Immediately post-brace application (power off), 3.Immediately post-brace activation (power on)
  To assess changes in basic walking speed over a short distance, reflecting potential improvements in mobility.
Surface Electromyography | 1.Baseline (before brace application) 2.Immediately post-brace application (power off), 3.Immediately post-brace activation (power on)
  To evaluate muscle activity patterns that indicate the orthosis's impact on muscle engagement during gait and sit to stand.
Gait Analysis | 1.Baseline (before brace application) 2.Immediately post-brace application (power off), 3.Immediately post-brace activation (power on)
  Using tools like the GAITRite system to obtain detailed measurements of gait cycle characteristics, providing comprehensive insights into the functional improvements afforded by the orthosis.

CONTACTS AND LOCATIONS:
Overall Officials: hyungik shin, prof, Principal Investigator — Seoul National University Hospital; Woo Hyung Lee, prof, Study Director — Seoul National University Hospital; Jung hyun Kim, prof, Study Director — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Jongno, South Korea

IPD SHARING:
Plan to Share IPD: No